CLINICAL TRIAL: NCT05739448
Title: Impact of an Intervention Combining Fortified Meals and Physical Activity in the Prevention of Undernutrition in Seniors : a Randomized Controlled Trial
Brief Title: Impact of an Intervention Combining Fortified Meals and Physical Activity in the Prevention of Undernutrition in Seniors
Acronym: FORTIPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAN WYMELBEKE ERA 2020
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Senior
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention)
- fortification (FOR) (Experimental)
  Interventions: Other: nutritional intervention
- fortification + physical activity (FAP) (Experimental)
  Interventions: Other: nutritional intervention; Other: physical activity

INTERVENTIONS:
Other: nutritional intervention — The nutritional intervention will be based on the following 4 elements: nutritional follow-up by a dietician, fortified meals, tender and juicy meat dishes and fish dishes
  Arms: fortification (FOR); fortification + physical activity (FAP)
Other: physical activity — The physical activity intervention will be based on the following 2 elements: Follow-up with a trainer for adapted exercise and physical exercise instruction sheets
  Arms: fortification + physical activity (FAP)

SUMMARY:
In the context of an aging population, preventing undernutrition and its associated risks in the elderly is a major challenge for the coming decade. Undernutrition, a recognized pathology of the elderly, has many negative impacts on the health and well-being of a person. It increases the risk of falls, fractures, pathological episodes and hospitalizations. It induces or aggravates a state of frailty and dependence, ultimately affecting the quality of life and life expectancy of the elderly.

A decline in appetite and insufficient food intake are key factors in the risk of undernutrition. Contrary to popular belief, energy and protein requirements do not decrease with age and are sometimes higher for the elderly than for younger people. However, several studies have shown that caloric and protein intakes are lower than recommended for the elderly. This decrease in appetite is also accompanied by a decrease in micronutrient intake. Inadequate micronutrient intakes are associated with the onset or more rapid progression of age-related diseases. For example, inadequate intakes of lipophilic micronutrients (carotenoids, fat-soluble vitamins A, D and E, long-chain omega-3 polyunsaturated fatty acids) are associated with a more rapid onset or worsening of age-related macular degeneration (AMD).

In order to prevent undernutrition, a major challenge is to allow elderly people with a poor appetite to cover their nutritional needs. Meal fortification, which consists of adding ingredients with high nutritional value to foods and beverages commonly consumed by the elderly, is a promising strategy. It allows for better adaptation to the preferences of the elderly, who are often reluctant to change their consumption habits. However, meal fortification remains largely unknown and underutilized. In parallel, several studies have shown that a high adherence to the Mediterranean diet, which is characterized by a high intake of these micronutrients, is associated with a 40% reduction in the risk of progression to AMD.

Finally, there is a strong link between physical activity and nutrition to prevent muscle wasting in the elderly. Indeed, the results show that an intervention combining protein supplementation and physical exercise has a greater effect on muscle protein synthesis than protein supplementation alone. However, advancing age is frequently accompanied by a decrease in physical activity and an increase in sedentary lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Person over 70 years of age
* Person living at home or in a relative's home
* Person with low level of physical activity (no more than 30 minutes of exercise for at least 2 days per week)

Exclusion Criteria:

* Person with a prescription for an oral nutritional supplement
* Anyone with allergies or intolerances to foods/ingredients used in the fortified foods
* Anyone with an aversion to fish
* Anyone on a restrictive diet or vegan/vegetarian diet
* Persons on a texture modified diet (blended, pureed)
* Person requiring enteral or parenteral nutrition
* Person suffering from dysphagia
* Person in a wheelchair
* Persons on special diets (texture modified, enteral, parenteral)
* Person under legal protection (guardianship, trusteeship)
* Person under a legal protection measure
* A person who is incapable or unable to give consent
* Person who is not affiliated or not a beneficiary of a social security system
* Person in a period of exclusion from a previous study

Secondary exclusion criteria :

* Person who is malnourished (MNA Long-Form score < 17)
* Person with low cognitive abilities (MMSE < 20) without a caregiver
* Person with a BMI ≥ 35 kg/m2
* Person with balance disorders (Get up and Go test execution time > 20 seconds or time in unipodal balance < 5 seconds).
* Person suffering from an acute pathology that can influence the vital prognosis (cancer, renal failure with dialysis...)
* Person suffering from chronic neuropsychological disorders altering the decisional capacities without the help of a close relative.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 209 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Weight gain or loss | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France